CLINICAL TRIAL: NCT00481312
Title: A Prospective, Multi-centre, Randomised, Double-blind Comparison of Intravenous Dexmedetomidine With Midazolam for Continuous Sedation of Ventilated Patients in Intensive Care Unit
Brief Title: Dexmedetomidine Versus Midazolam for Continuous Sedation in the Intensive Care Unit (ICU)
Acronym: MIDEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3005013
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2009-11

CONDITIONS: Continuous Sedation in Initially Sedated Adults in ICU
Keywords: Initial Sedation; Mechanical ventilation
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- 2 (Active Comparator): Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Continuous Infusion
  Arms: 1
Drug: Midazolam — Continuous Infusion
  Arms: 2

SUMMARY:
Patients in ICU who need help with their breathing are put onto a machine called a ventilator and are also given a medicine, called a sedative, which helps them to sleep and makes them more comfortable. Midazolam is a sedative that is routinely used for these purposes.

For most patients the aim of sedation is to make them sleepy but still able to respond to nursing staff (light sedation)

Dexmedetomidine is a new sedative for use in intensive care and in this clinical study, dexmedetomidine is compared to midazolam. It is thought that dexmedetomidine might be slightly better at allowing patients to be sleepy but still respond to people around them. It also does not appear to affect patient's breathing. the purpose of this study is to test whether dexmedetomidine really does have these advantages compared to midazolam.

in this study we hope to show that: dexmedetomidine is at least as good as midazolam in helping patients to sleep better and making them more comfortable, and that they are able to co-operate better with the staff treating them, and that patients treated with dexmedetomidine require a shorter time on the ventilator than those treated with midazolam.

DETAILED DESCRIPTION:
This is a phase III, multi-centre, prospective, randomised, double-blind, double-dummy, active comparator study. The study consists of three periods: screening, double-dummy treatment and follow-up period.

All patients admitted to ICU will be pre-screened according to inclusion and exclusion criteria prior to informed consent using available clinical data.

Informed consent, screening and randomisation procedures should be completed within 72 hours from the time of admission to ICU and within 48 hours from starting continuous sedation. Eligible study subjects requiring light to moderate sedation (Richmond Agitation-Sedation Scale [RASS] = 0 to -3) will be randomised to either continue on midazolam or switch to dexmedetomidine. Patients should not have received any other continuously or regularly administered sedative agent than midazolam infusion during the last 12 hours except for opioid analgesics. Study treatments will be titrated to achieve an individually targeted sedation range determined on a daily basis. Rescue treatment (i.e. propofol boli) may be given if needed to achieve the target depth of sedation. Continued need for sedation will be assessed at a daily sedation stop, conducted at the same time each day. First sedation stop may be 12-36 hours from randomisation, depending on the time of day the study subject is randomised. The duration of study treatment is limited to a maximum of 14 days from randomisation. Following withdrawal of sedation, study subjects will be monitored for 48 hours and contacted by telephone 31 and 45 days after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Clinical need for sedation of an initially intubated (or tracheotomised) and ventilated (with inspiratory assistance) patient
* Prescribed light to moderate sedation (target RASS = 0 to -3) using midazolam infusion
* Patients should be randomised within 72 hours from ICU admission and within 48 hours of commencing continuous sedation in the ICU
* Patients should have an expected requirement for sedation of at least 24 hours from time of randomisation
* Written informed consent must be obtained according to local regulations before starting any study procedures other than pre-screening.

Exclusion Criteria:

* Acute severe intracranial or spinal neurological disorder due to vascular causes, infection, intracranial expansion or injury
* Uncompensated acute circulatory failure at time of randomisation (severe hypotension with MAP < 55 mmHg despite volume and pressors)
* Severe bradycardia (HR < 50 beats/min)
* AV-conduction block II-III (unless pacemaker installed)
* Severe hepatic impairment (bilirubin > 101 µmol/L)
* Need for muscle relaxation at the time of randomisation (may only be used for intubation and initial stabilization)
* Loss of hearing or vision, or any other condition which would significantly interfere with the collection of study data
* Burn injuries requiring regular anaesthesia or surgery
* Use of centrally acting α2 agonists or antagonists at the time of randomisation, notably clonidine (see section 5.7 for prior and concomitant treatments)
* Known allergy to any of the study drugs or any excipients of the study drugs
* Patients who have or are expected to have treatment withdrawn or withheld due to poor prognosis
* Patients receiving sedation for therapeutic indications rather than to tolerate the ventilator (e.g. epilepsy)
* Patients unlikely to require continuous sedation during mechanical ventilation (e.g. Guillain-Barré syndrome)
* Patients who are unlikely to be weaned from mechanical ventilation; e.g. diseases/injuries primarily affecting the neuromuscular function of the respiratory apparatus such as clearly irreversible disease requiring prolonged ventilatory support (e.g. high spinal cord injury or advanced amyotrophic lateral sclerosis)
* Distal paraplegia
* Positive pregnancy test or currently lactating
* Received any investigational drug within the preceding 30 days
* Concurrent participation in any other interventional study (any study in which patients are allocated to different treatment groups and/or non-routine diagnostic or monitoring procedures are performed)
* Previous participation in this study
* Any other condition which, in the investigator's opinion, would make it detrimental for the subject to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Depth of sedation using the RASS. The target RASS range (target depth of sedation) should be 0 to -3 for a patient to be included in the study. The target may be amended during the study treatment, if clinically required | RASS score will be assessed approximately 2 hourly during the treatment period and during the 48-hour follow-up period
Duration of mechanical ventilation the number of days the patient receives mechanical ventilation will be recorded | This variable will be dependent on the individual patient and the number of days they require mechanical ventilation .

SECONDARY OUTCOMES:
Nurse's assessment of subject communication with visual analogue scales (VAS)Patients rousability and ability to co-operate and communicate will be measured using a visual analogue scale. | This will be measured at the end of every nursing shift whilst the patient remains on study treatment (maximum 14 days)
Length of ICU stay | Number of days a patient is in ICU which will vary depending on the underlying illness of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Jakob, MD PhD, Principal Investigator — Insel Spital, Bern CH-3010 Switzerland; Angela Ruck, BSc PhD, Study Director — Orion Pharma R&D Nottingham England
Locations (43):
- Belgium (4):
  - ULB Erasme, Route de Lennik, Brussels
  - UZ Brussel, Intensive Care Dept. Laarbeeklaan 101, Brussels
  - Universitaer Ziekenhuis Gent, Intensieve Zorgen, De Pintelaan 185, Ghent
  - CHU de Liege (Sart Tilman), Domaine de Sart-Tilman, Liège
- Estonia (4):
  - East Tallinn Central Hospital, Ravi Stret 18, Tallinn
  - North Estonian Regional Hospital, Centre of Intensive Care, J. Sutiste Tee 18, Tallinn
  - North Estonian Regional Hospital, Dept. of Postoperative Intensive Care, J. Sutiste Tee 18, Tallinn
  - Tartu University Hospistal, Clinic of Anesthesiology and Intensive Care, L. Puusepa 8, Tartu
- Finland (2):
  - Tampere University Hospital, ICU, Tampere, Pirkanmaa
  - Oulu University Hospital, Kajaanintie 50, Oulu
- France (12):
  - Centre Hospitalier Universitaire d'Angers, Reanimation medicale est de Mededicne Hyperbare, 4 Rue Larrey, Angers
  - Centre Hospitalier Victor Dupouy Hopital Dupuytren, Service Reanimation Polyvalente, 69, Rue du Lt Colonel Prud'hon, Argenteuil
  - Centre Hospitalier Universitaire de Grenoble, Service de Reanimation Medicale, Boulevard de la Chantourne, BP 217, Grenoble
  - Centre Hospitalier La Roche sur Yon CHD les Oudaireis, Service Reanimation CHD la Roche sur Yon, Les Oudairies, La Roche-sur-Yon
  - Hopital Albert Calmette, Boulevard Du Pr. Jules Leclercq, Lille
  - Centre Hospitalier Universitaire Limoges Hopital Dupuytren, Service de Reanimation Polyvalente, 2, Avenue Martin Luther King, Limoges
  - Centre Hospitalier Universitaire d'Orleans, Reanimation Medicale, 1, rue Prote Madeleine, BP 2439, Orléans
  - Hopital Bichat-Claude, Dept. D'Anasehesie et Reanimation Chirurgicale, 46, rue Henri-Huchard, Paris
  - Groupe Hospitalier Cochin Saint Vincent de Paul, Service de Reanimation Medicale, 27 Rue du Faubourg Saint Jacques, Paris
  - Hopital Foch, Service Renimation, 40 Rue Worth, Suresnes Hauts de Seine, Paris
  - Centre Hospitalier Universitaire de Poitiers, Reanimation Medicale, 2, Rue de la Miletrie, Poitiers
  - Centre Hospitalier Regional et Universitaire - Hopital Bretonneau Service Reanimation Medicale Polyvalente, 2, Boulevard Tonnelle, Tours cedex 9, Tours
- Germany (3):
  - Universitatsklinikum Bonn, Klinik u. Poliklinik f. Anasthesiologie u. Operative Intensivmedizin, Sigmund-Freud-Strasse 25, Bonn
  - Universitatsklinikum Greifswald, Klinik u. Poliklinik f. Anasthesiologie u. Intensivmedizin, Friedrich-Loeffler-Str. 23b, Greifswald
  - Universitatsklinikum Tubingen, Klinik fur Anasthesiologie und Intensivmedizin, Hoppe-Seyler-Strasse 3, Tübingen
- Netherlands (8):
  - VU Medisch Centrum, De Boelelaan 1117, Amsterdam
  - Gelre Hospitals - Locatie Lucas, A.Schweitzerlaan 32, Apeldoorn
  - Amphia Ziekenhuis, Dept. Intensieve Zorgen, Molengracht 21, Breda
  - Albert Schweitzer Hospital, Locatie Dordwikj, Albert Schweitzerplaats 25, Dordrecht
  - Kennemer Hospital, Boeerhaavelaan 29, Haarlem
  - Saint Elisabeth Ziekenhuis, Dept. Intensieve Zorgen, Hilvarenbeekseweg 60, Tilburg
  - Viecuri MC voor Noord-Limburg, Locatie Venlo, Dept. Intensieve Zorgen, Tegelseweg 210, Venlo
  - Isala Klinieken, Locatie Weezenlanden, Groot Wezenland 20, Zwolle
- Norway (4):
  - Haukeland University Hospital, Intensive Care Unit, Jonas Liesvei 65, Bergen
  - Rikshospitalet, Universitetsklinikk, Sognsvannsveien 20, Oslo
  - Ulleval University Hospital, Medical and Surgical ICU, Kirkeveien 166, Oslo
  - Aker Universtetssykehus HF, Anestesiavdelingen, Trondheimsveien 235, Oslo
- Switzerland (3):
  - Inselspital, Freiburgstrasse 4, Bern
  - Kantonsspital Winterthur, Brauerstrasse 15,, Winterthur
  - Universitatsspital Zurich, Klinik fur Innere Medizin, Intensivstation, Ramistrasse 100, Zurich
- United Kingdom (3):
  - University Hospital Birmingham, Department of Anaesthesia, Queen Elizabeth Hospital,, Birmingham
  - Birmingham Heartlands Hospital, Bordesely Green East, Birmingham
  - Derriford Hospital, Dept. of Intensive Care Level 4, Derriford Road, Plymouth

REFERENCES:
- [Derived] Turunen H, Jakob SM, Ruokonen E, Kaukonen KM, Sarapohja T, Apajasalo M, Takala J. Dexmedetomidine versus standard care sedation with propofol or midazolam in intensive care: an economic evaluation. Crit Care. 2015 Feb 19;19(1):67. doi: 10.1186/s13054-015-0787-y. PMID 25887576
- [Derived] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955